CLINICAL TRIAL: NCT03755193
Title: Examination of Efficacy and Safety of SERM or Bisphosphonates After 2-year-Denosumab Therapy in Japanese Osteoporosis Patients
Brief Title: Examination of Efficacy and Safety of Other Anti-Resorption Drugs After 2-year-Denosumab Therapy in Japanese Osteoporosis Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Lecturer at Shinshu University School of Medicine, Shinshu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DMAb switch 2018
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Diphosphonates

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SERM plus ELD (Active Comparator): To examine the effects of SERM plus ELD in osteoporosis patients
  Interventions: Drug: SERM "Viviant®Tablet 20mg" and ELD "Edirol®Tablet 0.75ug"; Drug: Bisphosphonates and ELD "Edirol®Tablet 0.75ug"; Drug: ELD "Edirol®Tablet 0.75ug"
- BP plus ELD (Active Comparator): To examine the effects of BP plus ELD in osteoporosis patients
  Interventions: Drug: SERM "Viviant®Tablet 20mg" and ELD "Edirol®Tablet 0.75ug"; Drug: Bisphosphonates and ELD "Edirol®Tablet 0.75ug"; Drug: ELD "Edirol®Tablet 0.75ug"
- ELD alone (Active Comparator): To examine the effects of ELD alone in osteoporosis patients
  Interventions: Drug: SERM "Viviant®Tablet 20mg" and ELD "Edirol®Tablet 0.75ug"; Drug: Bisphosphonates and ELD "Edirol®Tablet 0.75ug"; Drug: ELD "Edirol®Tablet 0.75ug"

INTERVENTIONS:
Drug: SERM "Viviant®Tablet 20mg" and ELD "Edirol®Tablet 0.75ug" — To examine the effects of SERM and ELD in osteoporosis patients
Drug: Bisphosphonates and ELD "Edirol®Tablet 0.75ug" — To examine the effects of BP and ELD in osteoporosis patients
Drug: ELD "Edirol®Tablet 0.75ug" — To examine the effects of ELD in osteoporosis patients

SUMMARY:
The aim of this study is to examine the efficacy and adverse events in the following 3 groups in Japanese osteoporosis patients after 2-year-denosumab therapy:

SERM and eldecalcitol treatment for 24 months Bisphosphonates and eldecalcitol treatment for 24 months Eldecalcitol treatment for 24 months

ELIGIBILITY:
Inclusion Criteria:

* osteoporosis patients

Exclusion Criteria:

* not osteoporosis patients who are allergic to the drugs, refused to do this research, or who are pregnant

Ages: 20 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-24 (Actual); Primary Completion 2024-11-23 (Estimated); Study Completion 2026-11-23 (Estimated)

PRIMARY OUTCOMES:
Assessment of bone mineral density in osteoporosis patients treated by SERM plus ELD, Bisphosphonate plus ELD, or ELD alone | Change from Baseline Values of bone mineral density at 2 years in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No